CLINICAL TRIAL: NCT02784717
Title: Xarelto® on Prevention of Stroke and Non-central Nervous System Systemic Embolism in Patients With Non-valvular Atrial Fibrillation in China: A Non-interventional Study
Brief Title: Xarelto on Prevention of Stroke and Non-central Nervous System Systemic Embolism in Patients With Non-valvular Atrial Fibrillation in China: A Non-interventional Study
Acronym: XASSURE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16819; XA1207CN (Other: Company internal)
Record Dates: First submitted 2016-04-27; First posted 2016-05-27 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: rivaroxaban,; non-interventional,; atrial fibrillation,; stroke prevention,
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban (Xarelto, BAY 59-7939): Female and male patients, who are at least 18 years of age with a diagnosis of non-valvular atrial fibrillation will be enrolled after the decision for a pharmacologic prophylaxis with rivaroxaban to prevent stroke or non-CNS systemic embolism has been made.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY 59-7939) — Decision regarding dose and duration of treatment made at the discretion of the attending investigator.

SUMMARY:
This non-interventional field study will investigate rivaroxaban under clinical practice conditions for stroke prevention and for prevention of non-CNS systemic embolism in patients with non-valvular atrial fibrillation in China.

DETAILED DESCRIPTION:
3000 patients will be provided with free drug.It is planned to have an interim analysis(IA) when 3000 patients are enrolled (cut off day is the 3000th patient completed at least 3 months follow-up visit). To end or continue enrolling patients will be decided based on the IA result and the evaluation comments from CFDA.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years of age diagnosed with non-valvular atrial fibrillation
* Patients for whom the decision to initiate treatment with rivaroxaban to prevent stroke or non-CNS systemic embolism was made as per investigator's routine treatment practice

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients, who are at least 18 years of age with a diagnosis of non-valvular atrial fibrillation will be enrolled after the decision for a pharmacologic prophylaxis with rivaroxaban within approved indication to prevent stroke or non-CNS systemic embolism has been made.
Sampling Method: Non-Probability Sample
Enrollment: 3055 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Number of Major bleeding events | Up to 30 months
  Major bleeding events, collected as serious or non serious adverse events and defined as overt bleeding associated with:
  1. a fall in haemoglobin of ≥2 g/dL, or
  2. a transfusion of ≥2 units of packed red blood cells or whole blood, or
  3. occurrence at a critical site (intracranial, intra-spinal, intraocular, pericardial, intra articular, intra-muscular with compartment syndrome, retroperitoneal), or
  4. death

SECONDARY OUTCOMES:
Number of Symptomatic thromboembolic events | Up to 30 months
  Collected as serious or non-serious adverse events
Number of Non-major bleeding | Up to 30 months
  Collected as serious or non-serious adverse events and defined as all bleeding events that do not fall in the category of major bleedings
Treatment satisfaction questionnaire | Up to 30 months
Adverse event and serious adverse event percentage in the different atrial fibrillation risk factor categories | Up to 30 months
Number of each reason for any switch from or interruption of rivaroxaban treatment | Up to 30 months
  If the patients switch from or interruption of rivaroxaban treatment, patients or physicians will be asked by several questions about the reasons of the switch and interruption, and collected in CRF. The reasons will be described by frequency distributions.
  Reason choice as below:
  1. Patient choice 2. Insufficient therapeutic effect 3. Adverse event 4. Surgery 5. Dentistry 6. Renal function change

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hangzhou, China

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/